CLINICAL TRIAL: NCT02777190
Title: A Comparison of Oral Misoprostol and Vaginal Misoprostol for Cervical Ripening and Induction of Labor
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient research staff to recruit and complete study
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Jaimey M. Pauli, MD, Principal Investigator, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00005107
Record Dates: First submitted 2016-05-17; First posted 2016-05-19 (Estimated); Results first posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Labor; Forced or Induced, Affecting Fetus or Newborn; Pregnancy
Keywords: misoprostol; cytotec; cervical ripening; labor, induced; active labor
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oral misoprostol (Experimental): oral misoprostol given 25 mcg every 2 hours
  Interventions: Drug: Misoprostol
- Vaginal misoprostol (Active Comparator): vaginal misoprostol given 25 mcg every 4 hours
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — Comparing dosing of misoprostol 25 mcg orally every 2 hours versus 25 mcg vaginally every 4 hours.
  Other Names: Cytotec

SUMMARY:
The purpose of this study is to study if misoprostol administered orally is at least as effective as misoprostol administered vaginally for cervical ripening and the induction of labor. The main purpose is to show that oral misoprostol administration is non-inferior to vaginal misoprostol administration with respect to the time interval from misoprostol administration to onset of active phase of labor. The study is a non-inferiority, prospective randomized controlled trial comparing oral misoprostol given as 25 mcg every 2 hours versus vaginal misoprostol given as 25 mcg every 4 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant Female Patients greater than or equal to 18 years of age
2. Induction of labor for a single live intrauterine pregnancy
3. Greater than or equal to 37 weeks gestational age
4. Cephalic presentation
5. 20 minute reassuring fetal heart rate (reactive nonstress test (NST))
6. Bishop score based on sterile vaginal exam of less than or equal to 6, for which the cervical dilation is less than or equal to 2 cm.
7. Equal to 3 or less uterine contractions over 10 minutes

Exclusion Criteria:

1. Previous uterine scar
2. Contraindication to vaginal delivery
3. Patients with preeclampsia
4. Grand multiparty - greater than or equal to 5 live births or stillbirths
5. Premature rupture of membranes
6. Suspected intrauterine growth restriction
7. Fetal anomalies
8. Contraindication to misoprostol (history of allergy to prostaglandins, glaucoma)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-04-23 (Actual); Study Completion 2019-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaimey Pauli, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kerr RS, Kumar N, Williams MJ, Cuthbert A, Aflaifel N, Haas DM, Weeks AD. Low-dose oral misoprostol for induction of labour. Cochrane Database Syst Rev. 2021 Jun 22;6(6):CD014484. doi: 10.1002/14651858.CD014484. PMID 34155622

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Misoprostol | Vaginal Misoprostol
Started | 17 | 17
Completed | 16 | 11
Not Completed | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Misoprostol | Vaginal Misoprostol | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.8 (4.3) | 26.5 (5.7) | 27.2 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 17 | 16 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 13 | 13 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Time to Active Labor
Description: Active phase of labor defined as greater than or equal to 6 cm cervical dilation
Time Frame: from start of induction of labor (first misoprostol administration) to active phase of labor, up to 3 days.
Population: Subjects who reached active phase of labor.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Oral Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 17 | 11
hours | 19.8 (10.6) | 21.4 (10.3)
Statistical Analysis 1: Comparison: Oral Misoprostol vs Vaginal Misoprostol; Test type: Non-Inferiority — Margin of 4 hours; p = 0.09, t-test, 1 sided; one-sided two-sample t-test with alpha=0.025; Mean Difference (Final Values) = -1.7, 97.5% CI 1-sided [upper limit 6.7] — Difference calculated as oral minus vaginal

2. Secondary Outcome: Time to Initiation of Oxytocin for Labor Augmentation
Description: The length of time (in hours) between the administration of misoprostol (first dose) and the first administration of oxytocin for labor augmentation.
Time Frame: From start of induction of labor (first misoprostol administration) to initiation of oxytocin for labor augmentation, up to 36 hours
Population: Subjects who initiated oxytocin
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Oral Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 15 | 15
hours | 11.0 (6.8) | 12.6 (6.8)
Statistical Analysis 1: Comparison: Oral Misoprostol vs Vaginal Misoprostol; Test type: Superiority; p = 0.54, t-test, 2 sided

3. Secondary Outcome: Time to Vaginal Delivery
Description: includes vaginal deliveries only; cesarean section deliveries are excluded
Time Frame: from start of induction of labor (first misoprostol administration) to vaginal delivery, up to 3 days
Population: vaginal deliveries
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Oral Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 15 | 10
hours | 22.3 (11.1) | 23.2 (9.7)
Statistical Analysis 1: Comparison: Oral Misoprostol vs Vaginal Misoprostol; Test type: Superiority; p = 0.64, t-test, 2 sided

4. Secondary Outcome: Cesarean Section Rate
Description: Number of cesarean sections/total deliveries (%)
Time Frame: From enrollment until delivery, up to 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 17 | 17
Participants | 2 | 7
Statistical Analysis 1: Comparison: Oral Misoprostol vs Vaginal Misoprostol; Test type: Superiority; p = 0.12, Fisher Exact

5. Secondary Outcome: Rate of Tachysystole
Description: Tachysystole is defined as 4 or more contractions in a 10 minute period.
Time Frame: from enrollment until delivery, up to 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 17 | 17
Participants | 1 | 4
Statistical Analysis 1: Comparison: Oral Misoprostol vs Vaginal Misoprostol; Test type: Superiority; p = 0.34, Fisher Exact

6. Secondary Outcome: Rate of Tachysystole Causing Non-reassuring Fetal Heart Tones
Description: Previously defined as "hyperstimulation", this outcome measure is defined as 4 or more contractions in a 10 minute period (tachysystole) thought to be causing recurrent variable or late decelerations, bradycardia, or minimal variability in the fetal heart rate tracing (non-reassuring fetal heart tones,which would require intervention to resolve or delivery of the infant).
Time Frame: From enrollment until delivery, up to 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 17 | 17
Participants | 1 | 2
Statistical Analysis 1: Comparison: Oral Misoprostol vs Vaginal Misoprostol; Test type: Superiority; p = 1.00, Fisher Exact

7. Secondary Outcome: Rate of Need for Tocolysis
Description: Tocolysis is the administration of medication to decrease or stop contractions.
Time Frame: from enrollment until delivery, up to 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 17 | 16
Participants | 1 | 2
Statistical Analysis 1: Comparison: Oral Misoprostol vs Vaginal Misoprostol; Test type: Superiority; p = 0.60, Fisher Exact

8. Secondary Outcome: Rate of Chorioamnionitis
Description: Chorioamnionitis is defined as an intraamniotic infection.
Time Frame: from enrollment until delivery, up to 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 17 | 17
Participants | 0 | 0

9. Secondary Outcome: Rate of Meconium Stained Fluid
Description: Amniotic fluid with visible meconium (from fetal defecation) within it.
Time Frame: from enrollment until delivery, up to 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 17 | 16
Participants | 2 | 4
Statistical Analysis 1: Comparison: Oral Misoprostol vs Vaginal Misoprostol; Test type: Superiority; p = 0.40, Fisher Exact

10. Secondary Outcome: Neonatal Morbidity
Description: binary composite outcome defined as Apgar score < 7, or cord blood gas pH of less than 7 or base deficit great than 12, or neonatal intensive care unit admission within 4 hours of delivery.
Time Frame: 4 hours from delivery
Population: Excludes neonates with APGAR score>7 not admitted to NICU but were missing cord blood gas results
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 10 | 12
Participants | 2 | 3
Statistical Analysis 1: Comparison: Oral Misoprostol vs Vaginal Misoprostol; Test type: Superiority; p = 1.00, Fisher Exact

11. Secondary Outcome: Rate of Anti-emetic Use
Description: Use of medication to treat nausea.
Time Frame: from enrollment until delivery, up to 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 17 | 17
Participants | 7 | 1
Statistical Analysis 1: Comparison: Oral Misoprostol vs Vaginal Misoprostol; Test type: Superiority; p = 0.04, Fisher Exact

12. Secondary Outcome: Rate of Vaginal Delivery Within 24 Hours
Description: Vaginal delivery within from start of induction with misoprostol.
Time Frame: 24 hours from start of induction of labor (first misoprostol administration)
Population: vaginal deliveries only
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 15 | 10
Participants | 10 | 6
Statistical Analysis 1: Comparison: Oral Misoprostol vs Vaginal Misoprostol; Test type: Superiority; p = 1.00, Fisher Exact

13. Secondary Outcome: Rate of Abandoning Misoprostol for Cervical Ripening and Switching to Mechanical Dilation for Cervical Ripening
Description: Based on clinician's judgment on the progress of the induction, the rate that misoprostol administration was stopped and a cervical ripening balloon was used instead
Time Frame: from enrollment until delivery, up to 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Misoprostol | Vaginal Misoprostol
Number analyzed (Participants) | 17 | 17
Participants | 2 | 7
Statistical Analysis 1: Comparison: Oral Misoprostol vs Vaginal Misoprostol; Test type: Superiority; p = 0.12, Fisher Exact

ADVERSE EVENTS:
Time Frame: During hospital stay-admission for induction until discharge after delivery, up to 7 days.
Description: Charts were reviewed for the specific events of postpartum hemorrhage requiring blood transfusion, maternal surgical ICU admission and neonatal NICU admission during the maternal hospital stay (admission for induction until discharge after delivery, up to 7 days).
Arm/Group | Oral Misoprostol | Vaginal Misoprostol
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 1/17 | 1/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Misoprostol (N=17) | Vaginal Misoprostol (N=17)
Neonatal NICU admission (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations include that during the COVID-19 pandemic, all in person research was suspended. Research time was reallocated to clinical time for providers. Recruitment was difficult. We had multiple changes in the research team requiring retraining. Ultimately, we were not able to recruit the numbers needed so the trial was terminated with inadequate numbers of subjects analyzed. Multiple turnovers led to a delay in completing our close out.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-09-15): https://cdn.clinicaltrials.gov/large-docs/90/NCT02777190/Prot_SAP_ICF_001.pdf